CLINICAL TRIAL: NCT01636362
Title: An Open, Non Controlled, Multi-centre, Clinical Investigation to Evaluate Efficacy in Partial Thickness (Superficial, Deep and Mixed) Second Degree Burns When Using a Soft Silicone, Silver Containing, Wound Contact Layer, Mepitel Ag.
Brief Title: A Clinical Investigation to Evaluate Efficacy of Mepitel Ag in Partial Thickness Second Degree Burns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MpT Ag 01
Record Dates: First submitted 2012-06-26; First posted 2012-07-10 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2013-12

CONDITIONS: Burns; Wound Healing
Keywords: Partial-thickness second degree burns; Mepitel Ag; Silver dressing
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mepitel Ag (Experimental): Mepitel Ag is an antimicrobial, meshed, non-adherent wound contact layer allowing passage of exudate and providing fixation and protection of tissues.
  Interventions: Device: Mepitel Ag

INTERVENTIONS:
Device: Mepitel Ag — Mepitel Ag is an antimicrobial, meshed, non-adherent wound contact layer allowing passage of exudate and providing fixation and protection of tissues.

SUMMARY:
Approximately 55-65 subjects from 3-6 sites suffering from a burn injury covering 1-25% Total Body Surface Area (TBSA) will be evaluated providing they fulfill all inclusion and none of the exclusion criteria and have given a signed and dated informed consent. Study site will be from 1-15%. Each subject will be followed once a week for a maximum of 3 weeks or until the burn is healed if that occurs earlier. All dressing changes will be performed at the clinic and gauze rolls will be used as secondary dressing. All dressing changes will be registered in a dressing log. All subjects will be consecutively allocated to a subject code.

DETAILED DESCRIPTION:
see Brief summary

ELIGIBILITY:
Inclusion Criteria:

* Subject with a partial-thickness (superficial, deep or mixed) second degree burn from 1-25% TBSA
* Study site is from 1-15% BSA
* Study site is a single, isolated burn area
* From 2 years and above
* Thermal burn injury
* Signed Informed Consent/Assent Form
* Subjects who are younger than the legal consenting age must in addition to their own Assent form have a signature from a legally authorized representative.

Exclusion Criteria:

* Completely non-exuding or dry wound bed at study site
* Full thickness >5%
* Burn greater than 24 hrs old
* Burns to face or neck
* Suspicion of infection of study burn
* Use of chemical/enzymatic and biological debridement within 7 days of investigation start
* Chronic steroid use, hx of skin malignancy or chronic papulosquamous disease (e.g. eczema, Pemphigus) and hx of Steven Johnson or TENS disease
* Subject with lung injury or subject being on a ventilator
* Subject with dermatologic skin disorders or necrotizing processes
* Subject with insulin dependent diabetes mellitus
* Electrical, chemical etiology
* Diagnosed underlying disease(s) (e.g. HIV/AIDS, cancer and severe anaemia), judged by the investigator to be a potential interference in the treatment
* Non-compliant subject
* Subject previously included in this investigation
* Subject included in other ongoing clinical investigation at present or during the past 30 days.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Silverstein, MD, Principal Investigator — INTEGRIS Baptist Medical Center, Inc. Paul Silverstein Burn Center
Locations (6):
- United States (6):
  - Arizona Burn Center, Phoenix, Arizona
  - Orlando Regional Medical Center, Orlando, Florida
  - Wishard, Indianapolis, Indiana
  - Paul Silverstein, MD, Oklahoma City, Oklahoma
  - S:t Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Harborview Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mepitel Ag
Started | 45
Completed | 37
Not Completed | 8
Not completed — Physician Decision | 6
Not completed — Subject healed, not returning | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Mepitel Ag
Number analyzed (Participants) | 45
Age, Continuous [Mean (Full Range); unit: years] | 25 [2 to 82]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17
  Between 18 and 65 years | 27
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Healed at Day 14.
Description: > = 95 % epitheliazation
Time Frame: Healing will be assessed after 14 days.
Measure: Number; unit: participants
Arm/Group | Mepitel Ag
Number analyzed (Participants) | 45
participants | 35

2. Primary Outcome: Proportion of Subjects Healed at Day 21.
Description: The proportion of subjects healed will be assessed at day 14. Wounds not healed at day 14 will be assessed again at day 21.
Time Frame: Healing will be assessed after 21 days.
Measure: Number; unit: participants
Arm/Group | Mepitel Ag
Number analyzed (Participants) | 37
participants | 37

3. Secondary Outcome: Percent of Study Burn Healed.
Description: Percent of study burn healed measured by PictZar photo analysis of tissue types.
Time Frame: At day 21
Measure: Median (Full Range); unit: percentage of healing
Arm/Group | Mepitel Ag
Number analyzed (Participants) | 37
percentage of healing | 97.1 (7,1) [75.6 to 100]

ADVERSE EVENTS:
Arm/Group | Mepitel Ag
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 3/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepitel Ag (N=45)
Increased pain (Skin and subcutaneous tissue disorders) | 1 (1) — # Increased burn pain, subject was seen one day early at the burn clinic. The study site was at that time healed. All burns were treated with Mepitel Ag.
Suspected cellulitis (Infections and infestations) | 1 (1) — # Suspected cellulitis
Increased pain (Skin and subcutaneous tissue disorders) | 1 (1) — Increased pain to RUE (right upper extremity), withdrawn from the investigation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other